CLINICAL TRIAL: NCT01662713
Title: Optical Frequency Domain Imaging for Non-melanoma Skin Cancers
Acronym: OFDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Benjamin Vakoc, Assistant Professor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2012P002430
Record Dates: First submitted 2012-08-08; First posted 2012-08-10 (Estimated); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Non-Melanoma Skin Cancer (NMSC)
Keywords: skin cancer; optical imaging; optical coherence tomography; optical frequency domain imaging
MeSH Terms: conditions — Skin Neoplasms | interventions — Optical Imaging; Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NMSC Imaging (Experimental): Optical Frequency Domain Imaging (OFDI) will be used to look at non melanoma skin cancer (NMSC) lesion(s).
  Interventions: Device: OFDI

INTERVENTIONS:
Device: OFDI — Imaging of skin
  Other Names: Optical Imaging; Optical Coherence Tomography; OCT; Optical Frequency Domain Imaging

SUMMARY:
The purpose of this research study is to find out if a non-invasive imaging device called Optical Frequency Domain Imaging (OFDI) can help doctors to see the tissue and blood vessels that are related to non-melanoma skin cancers. OFDI was designed to see microscopic details of your skin without needing to use any invasive techniques such as surgery or biopsy.

DETAILED DESCRIPTION:
Non-melanoma skin cancer (NMSC) is the most common cancer in the United States, with more than 750,000 diagnosed patients treated every year. Its prevalence and incidence have significantly increased over the past two decades and it has been estimated that 20% of all Americans will develop this type of cancer during their lifetime (Neville et al., 2007). Biopsy and surgical resection of NMSC can result in tissue mutilation and scaring. Therefore, there is a need for new imaging technologies that can be used to non-invasively guide biopsy and surgery.

Optical Frequency Domain Imaging (OFDI) is a second-generation imaging implementation of optical coherence tomography (OCT) developed at the Wellman Center. OFDI provides high-resolution three-dimensional imaging in tissue. It uses an interferometric depth-sectioning technique and employs a near-infrared light source. Through analysis of phase information in the recorded signal. OFDI can detect blood vessels within tissues and tumors. Importantly, OFDI-based vascular imaging can be performed without the need for exogenous contrast agents, making it relatively easy to deploy in clinical settings.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects with Fitzpatrick skin type I-VI
2. Subjects with ages between 18 and 80 years of age
3. Presence of at least one NMSC lesion

Exclusion Criteria:

1. Subjects with active localized or systemic infections
2. Subjects participating in potentially confounding clinical studies of investigational therapies, either drug or device.
3. Subjects taking any topical/systemic chemotherapy or immunosuppressants
4. Subjects who are pregnant and/or breastfeeding
5. Subjects with tape adhesive allergies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Successful imaging of lesion | After completion of imaging session
  Images acquired of NMSC

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Vakoc, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States